CLINICAL TRIAL: NCT00933881
Title: A Pilot Study to Evaluate the Association Between Gestational Diabetes, Heart Rate Variability and Sleep-Disordered Breathing
Brief Title: Gestational Diabetes and Sleep-Disordered Breathing
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: 28143
Record Dates: First submitted 2009-07-06; First posted 2009-07-07 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Gestational Diabetes Mellitus
Keywords: GDM
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gestational Diabetes Mellitus (GDM)
  Interventions: Other: Determining a change in heart rate variability post delivery of the baby

INTERVENTIONS:
Other: Determining a change in heart rate variability post delivery of the baby — Determining a change in heart rate variability post delivery of the baby

SUMMARY:
This study is designed to evaluate the amount of heart rate variability (HRV) for women with gestational diabetes mellitus (GDM) and to determine whether women with GDM have transient sleep-disordered breathing (SDB) during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women aged 18-40 years old.
2. Pregnant women at gestational age 30 to 34 weeks.

Exclusion Criteria:

1. Pregnant women with known type 1 or type 2 diabetes mellitus.
2. Pregnant women carrying more than one fetus.
3. Pregnant women with pre-gestational hypertension.
4. Pregnant women with pre-eclampsia during current pregnancy.
5. Pregnant women with a history of coronary artery disease or acute ischemia.
6. Pregnant women who currently smoke.
7. Pregnant women without results for the 3 hour 100 gram oral glucose tolerance test.
8. Pregnant women with preterm labor, cervical shortening, premature rupture of membranes or any other obstetric complications that may predispose to preterm labor.
9. Pregnant women using 17-P (progesterone) to prevent recurrent pre-term labor.
10. Pregnant women with known SDB.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with Gestational Diabetes Mellitus (GDM)
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Improvement in heart rate control post-GDM | Two months after delivery

SECONDARY OUTCOMES:
Improvement in SDB post-GDM | Two months after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Christiana Care Health Services, Newark, Delaware, United States